CLINICAL TRIAL: NCT03015610
Title: Genotype-tailored Treatment of Symptomatic Acid-Reflux in Children With Uncontrolled Asthma
Acronym: GenARA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Lang, M.D., M.P.H. (Other)
Collaborators: Thrasher Research Fund (Other); Nemours Children's Clinic (Other)
Responsible Party: Sponsor-Investigator, Jason Lang, M.D., M.P.H., Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00079073
Record Dates: First submitted 2016-12-13; First posted 2017-01-10 (Estimated); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Gastroesophageal Reflux
Keywords: Personalized Medicine; CYP2C19; Lansoprazole; Pharmacokinetics
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): participants will receive oral blinded matched placebo once daily
  Interventions: Drug: matched placebo
- Genotype-guided Lansoprazole (Experimental): participants will receive oral blinded commercially available lansoprazole once daily with a dose appropriate for the participant's metabolizer phenotype
  Interventions: Drug: commercially available lansoprazole

INTERVENTIONS:
Drug: commercially available lansoprazole — these participants will receive a one-time dose of lansoprazole followed by PK analysis and then once daily lansoprazole for 24 weeks
  Other Names: once daily
  Arms: Genotype-guided Lansoprazole
Drug: matched placebo — these participants will receive a one-time dose of lansoprazole followed by PK analysis and then once daily placebo for 24 weeks
  Other Names: once daily
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of CYP2C19 and ABCB1 genes on pharmacokinetics of lansoprazole in children with mild gastroesophageal reflux (GER) and uncontrolled asthma. It will determine if genotype-guided lansoprazole dosing of lansoprazole improves GER and asthma control.

DETAILED DESCRIPTION:
BACKGROUND: Poorly controlled asthma especially in children remains a major public health problem. Many children with poor asthma control experience gastroesophageal reflux (GERD). The effect of mild GERD on asthma remains controversial despite studies involving proton-pump inhibitors (PPIs) assessing their effect on asthma. Past inconsistent findings regarding the effect of PPIs on asthma control may have resulted from ineffective dosing strategies of proton-pump inhibitors employed in these studies. Drug levels and efficacy vary widely in the population and depend on genetics. Dosing in children which adjusts for the gene CYP2C19 may improve efficacy and reduce side-effects leading to improved asthma control.

HYPOTHESIS: #1: The investigators hypothesize that genotype-tailored lansoprazole dosing will reduce asthma symptoms in children with mild symptoms of GERD compared to placebo. #2: CYP2C19 and ABCB1 genetic variants influence the pharmacokinetics (drug levels) of lansoprazole as determined by population pharmacokinetic modeling.

METHODS: The investigators will conduct a 6-month randomized controlled trial comparing genotype-tailored lansoprazole dosing versus matched placebo in the control of asthma symptoms in 6-17 year olds with asthma and mild reflux. All participants will have baseline pharmacokinetics analysis following a single genotype-tailored dose to assess the effects of CYP2C19 and ABCB1.

IMPACT: These results would be a major advance in the science of safe dosing of proton-pump inhibitors in children and for the management of the millions of children struggling with reflux and asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-17 year olds with documented clinician-diagnosed asthma
* Evidence of recent uncontrolled asthma (must meet at least one of the following). This convention for defining poorly-controlled asthma has been successfully used in a large pediatric trial.

  * ACQ > 1.2
  * Use of short-acting beta-agonist for asthma symptoms twice/week or more on average over the past month
  * Nocturnal awakenings with asthma symptoms more than once per week on average over the last month
  * Two or more emergency department visits, unscheduled provider visits, prednisone courses or hospitalizations for asthma in the past 12 months
* Currently on stable dose of daily inhaled corticosteroid medication (ICS) for asthma control equivalent to 88mcg of fluticasone or greater for at least 6 weeks from the time of enrollment. Participant must be on National Asthma Education and Prevention Program (NAEPP) controller step 2, 3 or 4.
* Currently with mild GERD symptoms reported at V1 defined by a score on the Pediatric GERD Symptom Assessment Score greater than 15 and less than 80. GSAS ranges from 0 to >440.

Exclusion Criteria:

* Taking daily CYP2C19 substrates, inducers or inhibitors medication
* Past or current history of moderate-severe GERD or related disorders (erosive esophagitis, peptic ulcer disease, eosinophilic esophagitis) which in the opinion of the pediatric gastroenterology safety specialist/study physician requires treatment with acid-blocking agents;
* Daily use of a PPI for more than 4 consecutive weeks in the past 6 months;
* previous intubation for asthma,
* admission to intensive care unit for more than 24 hours for asthma in the past year,
* Previous surgery involving the esophagus or stomach (anti-reflux surgery, peptic ulcer surgery, trachea-esophageal fistula repair);
* Forced expiratory volume in 1 second (FEV1) < 60% of predicted at enrollment;
* Any major chronic illness that would interfere with participation in the intervention or completion of the study procedures;
* History of phenylketonuria (PKU);
* Medication use: treatment of GERD symptoms with over-the-counter antacids 4 days/week or more on average over past month;
* Theophylline preparations, azoles, anti-coagulants, insulin for Type 1 diabetes, digitalis, oral iron supplements when administered for iron deficiency within 1 month;
* Any investigational drugs within the past 2 months;
* Drug Allergies: previous allergic reaction from lansoprazole or other proton pump inhibitor medication or adverse reaction to aspartame;
* Inability to complete baseline measurements in a satisfactory manner according to the judgment of the research coordinator or site PI;
* Less than 75% completion of daily diary for asthma symptoms, SABA use and ICS medication adherence during the run-in period;
* Plan for family to move from study location within the next 6 months.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Lang, MD, MPH, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Nemours Children's Specialty Care, Jacksonville, Florida
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Genotype-guided Lansoprazole
Started | 17 | 18
Completed | 16 | 13
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Genotype-guided Lansoprazole | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (3.6) | 10.8 (3.3) | 10.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 6 | 4 | 10
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Questionnaire (ACQ) From Screening Through Week 26
Description: The ACQ considers a broad set of common indicators of asthma control including use of bronchodilators, cough, nocturnal symptoms, level of activity, and pulmonary function. Scores range between 0 (totally controlled) and 6 (severely uncontrolled). Reported is the change from week 0 to week 26; a negative change value indicates an improvement in asthma control.
Time Frame: Week 0 (baseline) to week 26
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 15 | 13
score on a scale | -0.5 (0.5) | -0.6 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.8716, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in GERD (Gastroesophageal Reflux Disease) Symptom Assessment Questionnaire Score (GSAS) From Screening Through Week 26
Description: A 10-item tool that has been validated in children in the assessment of gastroesophageal reflux disease related symptoms such as chest/abdominal pain, pain/choking with eating, swallowing dysfunction, regurgitation and nausea. It assesses symptom frequency and severity from the previous 7-days on an 8-point scale with 0 and 7 indicating the least and greatest severity, respectively. The total score ranges from 0 to 70, where a higher score indicates greater GERD symptom severity. Reported is the change from week 0 to week 26.
Time Frame: Week 0 (baseline) to week 26
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 15 | 14
score on a scale | -32.3 (18.7) | 23.4 (21.4)
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.2471, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Asthma Symptom Utility Index (ASUI) From Screening Through Week 26
Description: Questionnaire measures changes in asthma control. Each of the 11 items are scored on a 4-point Likert scale to assess frequency (not at all, 1 to 3 days, 4 to 7 days, and 8 to 14 days) and severity (not applicable, mild, moderate, and severe). The adjusted overall score ranges from 0 (worst possible symptoms) to 1 (no symptoms). Reported is the change from week 0 to week 26.
Time Frame: Week 0 (baseline) to week 26
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 12 | 9
score on a scale | 0 (0.2) | -0.1 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.039, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Annualized Rate of Asthma Exacerbations
Description: An exacerbation will be defined per the recommendations of the NIH Asthma Exacerbation Taskforce and will be defined as a worsening of asthma requiring the use of a systemic corticosteroid (at least 3 days of prednisolone/ prednisone or ≥1 days of dexamethasone) to prevent asthma worsening.
Time Frame: Up to week 26
Measure: Median (Inter-Quartile Range); unit: exacerbations per participant per year
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 17 | 18
exacerbations per participant per year | 0 [0 to 0] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.2765, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Annualized Rate of Episodes of Poor Asthma Control (EPAC)
Description: A study EPAC will be present if the participant meets any of the following criteria, (1) addition of systemic corticosteroid medication for asthma or (2) any unscheduled encounter to a non-study related health care provider (phone contact, ED, urgent care, hospital) for asthma symptoms.
Time Frame: Up to week 26
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 17 | 18
episodes per participant per year | 0 [0 to 0] | 0 [0 to 2.08]
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.191, Negative binomial regression; Risk Ratio (RR) = 2.32, 95% CI 2-sided [0.66 to 8.20]

6. Secondary Outcome: Annualized Rate of Respiratory Tract Infection (RTI)
Description: Participants/Caregivers will be asked to report diagnoses of RTI that occurred during the treatment period using interval reporting. RTI will include: (1) bronchitis, (2) otitis, (3) pneumonia.
Time Frame: Up to week 26
Measure: Median (Inter-Quartile Range); unit: RTIs per participant per year
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 17 | 18
RTIs per participant per year | 4.16 [2.26 to 12.0] | 4.0 [1.86 to 4.16]
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.0435, Negative binomial regression; Risk Ratio (RR) = 0.53, 95% CI 2-sided [0.29 to 0.98]

7. Secondary Outcome: Change in Lung Function Testing From Screening Through Week 26
Description: Forced Expiratory Volume in 1 Second (FEV1) measurement (mean change in FEV1 percent predicted from screening).
Time Frame: Week -2 (screening) to week 26
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Placebo | Genotype-guided Lansoprazole
Number analyzed (Participants) | 14 | 12
percentage of predicted value | 4.4 (16.1) | -3.7 (17.6)
Statistical Analysis 1: Comparison: Placebo vs Genotype-guided Lansoprazole; Test type: Superiority; p = 0.3808, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | Genotype-guided Lansoprazole
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 13/17 | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=17) | Genotype-guided Lansoprazole (N=18)
Headaches (Nervous system disorders) | 11 | 15
Nausea (Gastrointestinal disorders) | 8 | 9
Bloating (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 8 | 7
Constipation (Gastrointestinal disorders) | 8 | 3
Flatulence (Gastrointestinal disorders) | 11 | 10
Skin rash (Skin and subcutaneous tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03015610/Prot_SAP_000.pdf